# LEADING RESEARCH APPLIED RESEARCH UNIVERSITY OF ANDALAS CLUSTER RESEARCH PUBLICATION ACCELERATION OF PROFESSORS



RESEARCH SUB TOPIC: FOOD SECURITY, DRUG, AND HEALTH RESEARCH

SUB TOPIC: NUTRITION AND HEALTH

# **RESEARCH TITLE**

# EFFECTS OF DADIH FUNCTIONAL BREAD ON THE MICROBIOTA PROFILE OF PREGNANT WOMEN AND INFANT BIRTH WEIGHT INCREASE

BY:

# PROPOSING RESEARCHER:

Dr. HELMIZAR, SKM, M. BIOMED NIDN. 0010117309 Dr. AZRIMAIDALIZA, SKM, MKM Dr. FERDINAL FERRY, SpOG (K) Dr. FRIMA ELDA, SKM, MKM dr. ASRAWATI, M.BIOMED, SpA (K)

**Document Date: 02 January 2023** 

This research was conducted in several stages including the following:

# 1. Participant Flow

Based on the results of the research implementation, there were 88 respondents and a baseline was carried out and intervention was given (giving bread and curd vla for 3 months). The respondents were divided into two groups, namely intervention and control. The intervention group is the group that is given the treatment and the control group is the placebo group.



# a. Recruitment Details

This research began on May 9 2022 to August 30 2022 (baseline stage 1) and at the baseline stage 2 on September 20 2022 it was continued with intervention and ended in November 2022. The working area of the health centered is several selected health centered in Padang City according to the Locus Stunting in Padang City.

# b. Title Group

Group 1 respondents were intervention respondents

### c. Group Definition

The intervention group is the group that was given the treatment (bread and curd custard).

### 2. Baseline Characteristics

Based on the table below, the total number of respondents who were successfully baselined was 106 people, but after being reconfirmed and adjusting to the inclusion criteria, 18 respondents dropped out. For this reason, the total number of respondents who took part in the research (intervention) was 88 people. The sample respondents will be divided into two groups, namely the intervention group and the control group.

| Research sites | Date and time | Number of<br>Samples |
|---|---|---|
| Andalas Health Center | Wednesday/27 July 2022 | 16 |
| Nanggalo I health center | Thursday/28 July 2022 | 29 |
| Nanggalo II Public Health Center | Tuesday/ September 20, 2022 | 19 |
| Kuranji I Health Center | Monday/ September 19, 2022 | 19 |
| Kuranji II Health Center | Tuesday/ September 20, 2022 | 23 |
| | Total (Drop Out 18 respondents) | 106 |
| | Total of All Samples | 88 |

# a. Group Information

Respondent criteria in this study are; mothers with a gestational age of 12-20 weeks, in good health, willing to take part in the study with the stages of filling out questionnaires, collecting blood, and participating in the puskesmas to carry out ultrasound examinations, not moving before delivery, not suffering from certain diseases such as ( Tuberculosis, Diabetes Mellitus, Hypertension, History of Preeclampsia, or currently taking regular medication). As well as signing an informed consent, and willing to consume curd bread and vla until delivery.

# b. Title Group

Group 1 respondents were intervention respondents

## c. Group Definition

The intervention group is the group that was given the treatment (bread and curd custard).

# d. Baseline Analysis of Population Information (Overall Total Baseline)

The overall baseline is 106 people.

# e. Basic Measurement Information

The basic measurements for pregnant women include mother's ethnicity, mother's education, mother's occupation, mother's knowledge, family income, family members who smoke, mother's age, and gestational age. Basic measurements for newborns include birth weight, birth length, head circumference, chest circumference, and arm circumference.

### f. Basic Measurement Title

The average maternal weight before and after the intervention, and the average body mass index measurement before and after the intervention.

# g. Specific Measurements

Specific measurements such as the mother's weight before and after giving the intervention, measuring the body mass index before and after the intervention, as well as measuring the acceptability of bread and curd products.

## h. Respondent Age

Respondents' ages were women of reproductive age ranging from 18 to 45 years.

### i. Gender

The specified gender is female.

# j. Race and Ethnicity

Minangkabau specific race and ethnicity

## k. Measurement Type

The number of participants was 88 people.

# I. Dispersion measure

Complete

# m. Baseline Measurement Data

The data is in the form of numbers in the results table.

### n. Unit of Measurement

The basic unit of measurement for age is years, for education level are elementary school, junior high school, senior high school, and college.

# 3. Outcome Measures

### a. Outcome measures Information

Based on the research that has been done, the results obtained are the mother's weight gain, difference, and body beat as well as the length of the baby's body that was born.

### b. Outcome measures Type

The type of outcome measure is primary data.

## c. Outcome measures Title

The title of the outcome measures was the acceptability test for bread products and dadih sauce in the intervention and control groups, the differences in mean body weight and body mass index in the baseline,

intervention, and control groups, and the differences in outcome in weight and birth length of infants in the intervention and control groups.

### d. Outcome Measurement Time frame



# e. Title Group

Group 1 respondents were intervention respondents and group 2 respondents were control respondents.

# f. Group Description

The intervention group is the group that was given the treatment (bread and curd custard).

# g. Baseline Analysis of Population Information (Overall Number of Participant Analyzed)

The overall baseline is 106 people.

# h. Outcome Measurement Type

The type of measurement of the results is the average.

### i. Dispersion measure

Complete

### j. Outcome Measures Data

The outcome measure data is attached to the manuscript to be submitted.

# k. Unit of Measure

The unit for measuring mother's weight is Kilograms, for height is Centimeters, for measuring baby's weight is Grams, and body length is Centimeters.

# l. Statistical analysis

Statistical analysis used a randomized controlled trial (RCT) design and previously performed a data normality test using Kolmogorov Smirnov and using the T-Independent test. With a p-value <0.05.

# 4. Adverse Events

# a. All-cause mortality

No, There is'nt

# b. Serious adverse events

No, There is'nt

### c. Other adverse events

No, There is'nt

# d. Time frame



### e. The collation approach for the default table

No, There is'nt

# f. The total number affected by all causes of death

No, There is'nt

# g. Total At-Risk Number of Deaths from All Causes

No, There is'nt

## h. Total Number Affected by Each Serious Adverse Event

No, There is'nt

### i. Total At Risk for Serious Adverse Events

4 people

# j. Frequency Threshold for Reporting Other Unexpected Events (Excluding Serious)

No, There is'nt

# k. Total Number Affected by Other Unexpected Events (Excluding Serious) Above the Frequency Threshold.

No, There is'nt

# 1. Total At Risk for Other Unexpected Events (Excluding Serious)

No, There is'nt

# m. Term Unexpected Event

Pregnancy, Postpartum, and Perinatal.

# n. Collection Approach

No, There is'nt

### o. Bad event data

Number of participants affected : None Number of at-risk participants : None Number of occurrences : None

### 5. Limitations and Caveats

The obstacle in this study was that at the time of recruitment there were also many mothers who did not want to participate because they were afraid of taking blood and the reason was that their husbands did not allow it. Apart from that, the delivery of curd bread and vla is sometimes hampered by rainy weather. The distance between the respondent's house is far enough to be traveled every day. In addition, there are also mothers who

are getting bored and nauseous consuming bread, because they are experiencing a phase of nausea and vomiting. And mothers want more varied types of bread so they don't get bored. The condition of the product is because it does not use preservatives so it quickly becomes sour and smells. So that mothers do not want to eat it. Mother's health condition is also an obstacle, due to the rainy season, many mothers are sick so they don't have an appetite to eat and consume curd vla bread. Besides that,

# 6. Certain Agreements

Yes. Sponsor's Employee Principal Investigator

# 7. Results Point of Contact

Official Name or Title : Dr. Helmizar, SKM, M. Biomed

Organization Name : University of Andalas
Telephone : +62 812-6776-930
E-mail : helmizar@ph.unand.ac.id

# 8. Delayed Results

No, There is'nt